CLINICAL TRIAL: NCT01717183
Title: Assessment of the Efficacy and Safety of a New Wound Dressing in the Local Treatment of Diabetic Foot Ulcers: a Prospective, Randomised, Controlled, Double-blind, European Multicentre Clinical Trial
Brief Title: Assessment of the Efficacy and Safety of a New Wound Dressing in the Local Treatment of Diabetic Foot Ulcers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Laboratoires URGO (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FI-12-05-310 3113
Record Dates: First submitted 2012-10-26; First posted 2012-10-30 (Estimated); Last update posted 2014-04-11 (Estimated); Status verified 2014-04

CONDITIONS: Diabetic Foot Ulcer(s)
Keywords: Patient
MeSH Terms: conditions — Diabetic Foot

ARMS (2):
- URGO 310 3113 dressing - new (Experimental): flexible, conformable, non-adhesive and non-occlusive lipido-colloid matrix that does not adhere to the wound.
  Interventions: Device: Urgo 310 3113
- URGO 310 3113 dressing (Placebo Comparator): flexible, conformable, non-adhesive and non-occlusive lipido-colloid matrix that does not adhere to the wound.
  Interventions: Device: Placebo URGO 310 3113 dressing

INTERVENTIONS:
Device: Urgo 310 3113 — URGO 310 3113 dressing may be changed every 2 to 4 days, and left in place for up to 7 days, depending on the level of exudate and the wound condition
  Arms: URGO 310 3113 dressing - new
Device: Placebo URGO 310 3113 dressing
  Arms: URGO 310 3113 dressing

SUMMARY:
The main purpose of this trial is to demonstrate that the new dressing is more effective than the current dressing in the local treatment of chronic foot ulcers in diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female over 18 years old who has provided his/her written informed consent
* Patient covered by the French national insurance system
* Patient with Type 1 or Type 2 diabetes mellitus with glycated hemoglobi(HbA1c) levels ≤ 10% (assayed in the previous 3 months. If not available, this assay must be performed during the run-in period)
* Inpatient or outpatient who can be monitored by the same investigating team throughout the duration of the study
* Patient who agrees to wear the prescribed off-loading system every day, associated with the test dressing
* DFU with adequate arterial blood supply in the target limb DFU grade I-C or II-C as defined by the University of Texas Diabetic Wound Classification
* Neuropathy confirmed by loss of protective sensation to monofilament test (Semmes-Weinstein 5.07 monofilament)
* DFU located on the toe or on the lateral, dorsal or plantar side of the foot
* Target DFU surface area between 1 cm² and 30 cm², following debridement DFU duration between 1 and 24 months
* No local clinical infection (as defined by IDSA/IWGDF criteria) for any wound (target DFU or not) on lower limbs
* DFU adequately debrided

Exclusion Criteria:

* Pregnant or breast-feeding woman or woman of childbearing potential not using effective means of contraception
* Patient who took part in another clinical trial in the previous month or who is to take part in another clinical trial in the 20 weeks following inclusion
* Patient with any known intolerance or allergy or reported adverse reaction to one of the components of the trial dressings
* Patient who has undergone surgery or surgical revascularization (vascular reconstruction or angioplasty) in the previous 2 months
* Patient who has presented an acute ischemic event (Acute Myocardial Infarction (AMI) or stroke) in the 3 months before inclusion
* Patient with Severe kidney failure, defined as requirement for dialysis
* Patient with a systemic infection not controlled by suitable antibiotic treatment
* Patient with known osteomyelitis
* Patient with leg ulcer(s), regardless of limb
* Patient with wounds other than the target DFU located on the heel or on the interdigital part of the foot
* Patient with an active neoplastic condition, treated by radiotherapy, chemotherapy, hormone therapy or immunosuppressant agents
* Patient treated for a chronic disease requiring high doses of systemic corticosteroids (≥ 40 mg.d-1 of prednisolone or equivalent)
* Patient with a severe illness that might lead to premature withdrawal from the trial
* DFU for which surgery or surgical revascularization is planned at any time during the study
* Deep DFU defined as stage III or IV (University of Texas Diabetic Wound Classification)
* DFU clinically infected as defined by IDSA/IWGDF criteria
* DFU with more than 20% of its surface area covered by black necrotic tissue following debridement
* DFU located on an amputation stump
* DFU with neoplastic component

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2013-04

PRIMARY OUTCOMES:
Percentage of complete wound closure

SECONDARY OUTCOMES:
Time to complete wound closure
Change in wound surface area

CONTACTS AND LOCATIONS:
Locations (1):
- Toulouse, France

REFERENCES:
- [Derived] Maunoury F, Oury A, Fortin S, Thomassin L, Bohbot S; Explorer Study. Cost-effectiveness of TLC-NOSF dressings versus neutral dressings for the treatment of diabetic foot ulcers in France. PLoS One. 2021 Jan 22;16(1):e0245652. doi: 10.1371/journal.pone.0245652. eCollection 2021. PMID 33481840
- [Derived] Edmonds M, Lazaro-Martinez JL, Alfayate-Garcia JM, Martini J, Petit JM, Rayman G, Lobmann R, Uccioli L, Sauvadet A, Bohbot S, Kerihuel JC, Piaggesi A. Sucrose octasulfate dressing versus control dressing in patients with neuroischaemic diabetic foot ulcers (Explorer): an international, multicentre, double-blind, randomised, controlled trial. Lancet Diabetes Endocrinol. 2018 Mar;6(3):186-196. doi: 10.1016/S2213-8587(17)30438-2. Epub 2017 Dec 20. PMID 29275068